CLINICAL TRIAL: NCT06989333
Title: A Single-arm Clinical Study of Local Spraying of GM-CSF Via Bronchoscopy in the Treatment of Autoimmune Pulmonary Alveolar Proteinosis
Brief Title: Local Spraying of GM-CSF Via Bronchoscopy in the Treatment of Autoimmune Pulmonary Alveolar Proteinosis
Acronym: aPAP and GMCSF
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiuwu Bai (Other)
Responsible Party: Sponsor-Investigator, Jiuwu Bai, associate chief physician, Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025051795
Record Dates: First submitted 2025-05-17; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Alveolar Proteinosis
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spraying GM-CSF (Experimental)
  Interventions: Drug: GM-CSF (granulocyte-macrophage colony-stimulating factor)

INTERVENTIONS:
Drug: GM-CSF (granulocyte-macrophage colony-stimulating factor) — Bronchoscopy under general anesthesia or sedation; The predetermined dose of recombinant GM-CSF was dissolved in normal saline. The diseased lung segments were located through bronchoscopy and the liquid medicine was sprayed.

SUMMARY:
This study aims to explore a new therapeutic approach: the feasibility, safety and preliminary efficacy of directly spraying GM-CSF into the airway through bronchoscopy for the treatment of aPAP.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 60 years old;
2. A clear diagnosis of aPAP must meet at least one of the following diagnostic criteria:

1) BALF appears "milky white"; Or cytological examination reveals a large amount of PAS-positive protein deposition; 2) HRCT shows typical "paving stone-like changes"; 3) Positive for serum GM-CSF antibody. 3. There are more than one of the following treatment indications: Symptoms such as progressive breathing difficulties, coughing, and shortness of breath after activity occur; 2) Without oxygen inhalation, PaO2 > 65 mmHg 3) Pulmonary function DLCO accounts for % of the predicted value, ranging from 60% to 80%, including the critical value.

4. No other PAP specific treatments (such as WLL, inhaled GM-CSF, biological agents, etc.) have been received recently (for more than 4 weeks).

5. Agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

1. Secondary PAP (such as secondary to blood diseases, etc.);
2. Patients with obvious pulmonary fibrosis, emphysema or irreversible lung function impairment;
3. Patients in the acute exacerbation stage;
4. Patients with other lung diseases (such as active pulmonary tuberculosis, bronchiectasis with purulent infection or other chronic infections; Have severe asthma, chronic bronchospasm, etc.
5. Have a history of allergy to GM-CSF antibodies or related drug components;
6. Patients who have participated in other clinical drug trials within the past three months;
7. Patients who have experienced severe complications related to bronchoscopy or are intolerant to bronchoscopy;
8. Concurrent with other serious cardiovascular and cerebrovascular diseases, hematological disorders, malignant tumors, etc.
9. Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Chest HRCT | 12 weeks

IPD SHARING:
Plan to Share IPD: No